CLINICAL TRIAL: NCT00837421
Title: The Ohio State University Sepsis Registry
Status: Terminated | Type: Observational
Why Stopped: Lack of resources has prevented the study from continuation.
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Naeem Ali, MD, Associate Professor, Ohio State University
Other Study IDs: 2005H0029
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Sepsis
Keywords: sepsis; registry
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- sepsis: sepsis survivors

SUMMARY:
Specific Aim #1: To collect follow-up information about patients with sepsis in the OSUMC MICU who survive to hospital discharge for future retrospective IRB-approved studies.

Specific Aim #2: To collect a registry of patients who would be interested in hearing more information about future prospective IRB-approved studies for survivors of sepsis.

Specific Aim #3: To collect a blood sample from patients with sepsis admitted to the OSUMC MICU for future retrospective IRB-approved studies.

DETAILED DESCRIPTION:
There are several goals of the Ohio State University Sepsis Registry and Blood Bank. First, we hope that, by collecting a cohort of patients with sepsis, we will provide information for future studies with data of specific relevance to sepsis (the Clinical Registry). Second, by following survivors of sepsis for a more prolonged period than prior studies, we will better understand the disease process and the duration of recovery (the Follow-up Registry). We will contact hospital survivors every six months to assess their vital status, living situation and employment. Furthermore, subjects will have the opportunity to find out about new studies as they arise. Finally, we will ask subjects for permission to collect a blood sample (10 cc) to use for future studies analyzing genetic and protein data. There will be a step-wise consent process that will allow subjects to opt out of any or all parts of the study.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to OSUMC MICU, ≥ 18 years, have consensus criteria for sepsis (infection plus two of four systemic inflammatory response syndrome [SIRS] signs [tachycardia, tachypnea, fever or hypothermia, leukocytosis or leukopenia]).

Exclusion Criteria:

* Consent not available or declined, prisoner, died before discharge (excluded from Follow-up Registry only), died before blood collected (excluded from Blood Bank only), onset of sepsis more than 24 hours prior to ICU admission. Patients who have sepsis onset more than 24 hours prior to ICU admission but spent the ENTIRETY of the current admission in the OSUMC ED will be eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospital intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2006-12; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
To collect follow-up information about patients with sepsis in the OSUMC MICU who survive to hospital discharge for future retrospective IRB-approved studies. | end of study

SECONDARY OUTCOMES:
To collect a blood sample from patients with sepsis admitted to the OSUMC MICU for future retrospective IRB-approved studies. | end of study

CONTACTS AND LOCATIONS:
Overall Officials: James M O'Brien, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
The study was terminated and after analysis data integrity issues prohibited accurate IPD sharing. The data records have been destroyed.